CLINICAL TRIAL: NCT01132573
Title: A Phase I Study of the Histone Deacetylase Inhibitor Entinostat (SNDX-275, NSC 706995) Plus Clofarabine for Philadelphia Chromosome-Negative, Poor Risk Acute Lymphoblastic Leukemia or Bilineage/Biphenotypic Leukemia in Newly Diagnosed Older Adults or in Adults With Relapsed and Refractory Disease
Brief Title: Entinostat and Clofarabine in Treating Patients With Newly Diagnosed, Relapsed, or Refractory Poor-Risk Acute Lymphoblastic Leukemia or Bilineage/Biphenotypic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01436; NCI-2011-01436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000671796; JHOC-MD017; J09112 (Other: Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center); 8298 (Other: CTEP); U01CA070095 (NIH); P30CA006973 (NIH)
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-04

CONDITIONS: Acute Leukemias of Ambiguous Lineage; Philadelphia Chromosome Negative Adult Precursor Acute Lymphoblastic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia; Untreated Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — entinostat; Clofarabine

ARMS (1):
- Treatment (entinostat and clofarabine) (Experimental): Patients receive entinostat PO on days 1 and 8 and clofarabine IV over 2 hours on days 3-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity (only for patients >= 60 years of age with newly diagnosed ALL or ABL who are unable or unwilling to tolerate standard multi-agent chemotherapy and patients with relapsed or refractory ALL or ABL).
  Patients 40-59 years of age with newly diagnosed ALL receive standard multi-agent induction chemotherapy beginning on day 11. Patients >= 21 years of age in their first relapse with sensitive disease begin initiation of allogeneic transplant after one course of entinostat and clofarabine.
  Interventions: Drug: entinostat; Drug: clofarabine; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: entinostat — Given PO
  Other Names: HDAC inhibitor SNDX-275; SNDX-275
Drug: clofarabine — Given IV
  Other Names: CAFdA; Clofarex; Clolar
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of entinostat when given together with clofarabine in treating patients with newly diagnosed, relapsed, or refractory poor-risk acute lymphoblastic leukemia or bilineage/biphenotypic leukemia. Entinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as clofarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving entinostat with clofarabine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility, tolerability, toxicities, and maximum tolerated dose (MTD) of entinostat plus clofarabine for: adult patients age 40 and over with newly diagnosed, poor-risk Philadelphia chromosome negative (Ph-) acute lymphoblastic leukemia (ALL) or bilineage/biphenotypic leukemia (ABL) prior to traditional cyclical multi-agent chemotherapy, and adults age 21 and over with relapsed or refractory ALL/ABL.

II. To determine if entinostat plus clofarabine can induce clinical responses in adults with newly diagnosed, poor-risk ALL/ABL and in adults with relapsed/refractory ALL/ABL.

SECONDARY OBJECTIVES:

I. To determine pharmacokinetics (PK) of entinostat alone and in combination with clofarabine.

II. To obtain descriptive preliminary pharmacodynamic (PD) data regarding the effects of entinostat alone and in combination with clofarabine on histone acetylation and global and gene specific methylation in leukemic blasts.

III. To obtain descriptive preliminary data regarding the effects of entinostat alone and in combination with clofarabine on deoxyribonucleic acid (DNA) damage and apoptosis in leukemic blasts and residual disease monitored by 6-color flow cytometry.

OUTLINE: This is a dose-escalation study of entinostat.

Patients receive entinostat orally (PO) on days 1 and 8 and clofarabine intravenously (IV) over 2 hours on days 3-7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity (only for patients at least 60 years of age with newly diagnosed ALL or ABL who are unable or unwilling to tolerate standard multi-agent chemotherapy and patients with relapsed or refractory ALL or ABL).

Patients 40-59 years of age with newly diagnosed ALL receive standard multi-agent induction chemotherapy beginning on day 11. Patients at least 21 years of age in their first relapse with sensitive disease begin initiation of allogeneic transplant after one course of entinostat and clofarabine.

After completion of study treatment, patients are followed up at 30, 60, 90, 180, and 360 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults age >= 40 years with the established, pathologically-confirmed diagnoses of newly diagnosed ALL or ABL are eligible for study; adults with relapsed and refractory ALL or ABL who are >= 21 years of age and who have progressive disease following their last therapy are eligible for study; the additional following criteria must be met:
* For adults with relapsed/refractory ALL, no more than 5 previous regimens
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Patients must be able to give informed consent
* Female patients of childbearing age must have negative pregnancy test
* Total white blood cell count (WBC) =< 150,000 with no evidence for ongoing or impending leukostasis
* Total bilirubin =< 2.0 mg/dL unless elevated due to Gilbert's disease, hemolysis or leukemic infiltration
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 × upper limit of normal (ULN) unless due to leukemic infiltration
* Serum creatinine =< 2.0 mg/dL
* Left ventricular ejection fraction (LVEF) >= 45% as measured by echocardiogram (ECHO) or multi gated acquisition (MUGA) scan
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 30 days after study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients who have undergone stem cell transplantation (SCT), autologous or allogeneic, are eligible provided that they are >= 4 weeks from stem cell infusion, have no active graft-vs-host disease (GVHD), and meet other eligibility criteria
* Patients who fail primary induction therapy or relapse after achieving complete remission (CR) are eligible if they have undergone no more than 5 prior cytotoxic regimen, >= 14 days off cytotoxic chemotherapy, and >= 2 weeks radiation therapy; patients must be off biologic therapies >= 7 days, must be off hematopoietic growth factors >= 3 days; if using hydroxyurea steroids, imatinib, arsenic, interferon, or other non-cytotoxics for blast count control, patient must be off for >= 24 hrs before starting entinostat plus clofarabine

Exclusion Criteria:

* Philadelphia chromosome positive ALL
* Patients may not have received previous treatment with entinostat or other histone deacetylase (HDAC) inhibitors (including valproic acid) or clofarabine within the previous 6 months
* Concomitant chemotherapy, radiation therapy, or immunotherapy
* Hyperleukocytosis with >= 150,000 blasts/uL (if using hydroxyurea, steroids, maintenance doses of 6-mercaptopurine and/or methotrexate, arsenic, interferon or leukapheresis for blast count control, patient must be off those agents for 24 hours prior to beginning entinostat plus clofarabine)
* Active disseminated intravascular coagulation (DIC)
* Active central nervous system (CNS) leukemia; patients with known previous CNS leukemia may continue to receive intrathecal therapy with cytarabine (ara-C), methotrexate, and/or thiotepa plus steroids as prophylaxis against reactivation of active CNS disease
* Use of investigational cytotoxic agents within 30 days or any anticancer therapy within 14 days before study entry, except for hydroxyurea and steroids, both of which must be discontinued at least 24 hours before study entry; the patient must have recovered from all acute toxicities from any previous therapy; the patient must have recovered from all acute toxicities from any previous therapy
* Patients must have discontinued all growth factors at least 3 days before study
* History of severe coronary artery disease, including myocardial infarction within the previous 3 months, arrhythmias other than atrial flutter or fibrillation requiring medication, or uncontrolled congestive heart failure
* Dyspnea at rest or with minimal exertion
* Active uncontrolled infection; patients with infection under active treatment and controlled with antibiotics are eligible
* Patients with active >= grade 2 graft versus host disease (GVHD)
* Presence of other life-threatening illness
* Patients with mental deficits and/or psychiatric history that preclude them from giving informed consent or from following protocol
* Pregnant or nursing women; breastfeeding should be discontinued if the mother is treated with entinostat
* Male and female patients who are fertile who do not agree to use an effective barrier method of birth control (i.e., hormonal or barrier method of birth control; abstinence) to avoid pregnancy during the study and for a minimum of 30 days after study treatment
* Previous history of or current seizure disorder
* Human immunodeficiency virus (HIV) infected patients who have cluster of differentiation (CD4) cell count =< 350/mm^3 or a history of acquired immunodeficiency syndrome (AIDS)-defining conditions

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-04; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Frequency of the observed toxicities based on the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 360 days
  The frequency of the observed toxicities will be tabulated by type and grade.
MTD of entinostat followed by clofarabine, defined as the dose at which less than 2 of 3 patients experience dose limiting toxicity graded according to NCI CTCAE version 4.0 | 21 days

SECONDARY OUTCOMES:
Percentage change in phosphorylated H2A histone family, member X (H2AX), an indication of DNA damage | From baseline to 360 days
  Will be evaluated as a continuous variable. Will be estimated including the 95% confidence interval.
Percentage change in apoptosis | From baseline to 360 days
  Will be estimated including the 95% confidence interval.
Percentage change in histone acetylation | From baseline to 360 days
  Will be estimated including the 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Gojo, Principal Investigator — Johns Hopkins University Sidney Kimmel Comprehensive Cancer Center
Locations (4):
- United States (4):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Colorado, Denver, Colorado
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland

REFERENCES:
- [Derived] Carraway HE, Sawalha Y, Gojo I, Lee MJ, Lee S, Tomita Y, Yuno A, Greer J, Smith BD, Pratz KW, Levis MJ, Gore SD, Ghosh N, Dezern A, Blackford AL, Baer MR, Gore L, Piekarz R, Trepel JB, Karp JE. Phase 1 study of the histone deacetylase inhibitor entinostat plus clofarabine for poor-risk Philadelphia chromosome-negative (newly diagnosed older adults or adults with relapsed refractory disease) acute lymphoblastic leukemia or biphenotypic leukemia. Leuk Res. 2021 Nov;110:106707. doi: 10.1016/j.leukres.2021.106707. Epub 2021 Sep 10. PMID 34563945